CLINICAL TRIAL: NCT03663205
Title: A Phase 3, Open-Label, Multicenter, Randomized Study to Investigate the Efficacy and Safety of Tislelizumab (BGB-A317) (Anti-PD1 Antibody) Combined With Platinum-Pemetrexed Versus Platinum-Pemetrexed Alone as First-line Treatment for Patients With Stage IIIB or IV Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Tislelizumab Versus Chemotherapy in Advanced Non-Squamous Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-304; CTR20180032 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2018-08-16; First posted 2018-09-10 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab + Platinum + Pemetrexed (Experimental): Tislelizumab 200 milligrams (mg) administered intravenously (IV) once every 3 weeks plus cisplatin 75 mg/m^2 or carboplatin area under the plasma or serum concentration-time curve (AUC) 5 once every 3 weeks for 4 to 6 cycles and pemetrexed 500 mg/m^2 once every 3 weeks until unacceptable toxicity or disease progression (each cycle is 21 days)
  Interventions: Drug: Tislelizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Platinum + Pemetrexed (Active Comparator): Cisplatin 75 mg/m^2 or carboplatin AUC 5 once every 3 weeks for 4 to 6 cycles and pemetrexed 500 mg/m^2 administered IV once every 3 weeks until unacceptable toxicity or disease progression (each cycle is 21 days)
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Tislelizumab — Administered intravenously
  Other Names: Tevimbra; BGB-A317
  Arms: Tislelizumab + Platinum + Pemetrexed
Drug: Cisplatin — Administered intravenously
Drug: Carboplatin — Administered intravenously
Drug: Pemetrexed — Administered intravenously

SUMMARY:
This study evaluated the efficacy and safety of tislelizumab in combination with platinum (cisplatin or carboplatin) and pemetrexed compared with platinum and pemetrexed alone as first-line treatment in participants with Stage IIIB or IV non-squamous non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, male or female, signed informed consent form
2. Advanced NSCLC diagnosed by pathological or clinical physicians
3. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 1
4. Participants must have ≥ 1 measurable lesion as defined per RECIST v1.1
5. Participants must have no prior systemic chemotherapy for advanced or metastatic NSCLC
6. Life expectancy ≥ 12 weeks
7. Participants must have adequate organ function
8. Male/female is willing to use a highly effective method of birth control

Exclusion Criteria:

1. Diagnosed with NSCLC but with epidermal growth factor receptor (EGFR)-sensitizing mutation or anaplastic lymphoma kinase (ALK) gene translocation
2. Received any approved systemic anticancer therapy within 28 days prior to the initiation of study treatment
3. Received prior treatment with EGFR inhibitors or ALK inhibitors
4. Received prior therapies targeting programmed cell death protein-1 (PD-1) or programmed cell death protein ligand-1 (PD-L1)
5. With history of interstitial lung disease, non-infectious pneumonitis or uncontrolled systemic diseases
6. Clinically significant pericardial effusion
7. Severe infections, active leptomeningeal disease or uncontrolled, untreated brain metastasis
8. Any major surgical procedure ≤ 28 days before randomization
9. Human immunodeficiency virus (HIV) infection
10. Participants with untreated hepatitis B or C virus (HBV/HCV)
11. Active autoimmune diseases or history of autoimmune diseases
12. History of allergic reactions to chemotherapy

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2023-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (47):
- China (47):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - The Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Changsha Central Hospital, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University Branch Shizi, Suzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Jinan Military General Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Hangzhou First Peoples Hospital, Hangzhou, Zhejiang
  - Zhejiang University College of Medicine Second Affiliated Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Lu S, Wang J, Yu Y, Yu X, Hu Y, Ai X, Ma Z, Li X, Zhuang W, Liu Y, Li W, Cui J, Wang D, Liao W, Zhou J, Wang Z, Sun Y, Qiu X, Gao J, Bao Y, Liang L, Wang M. Tislelizumab Plus Chemotherapy as First-Line Treatment for Locally Advanced or Metastatic Nonsquamous NSCLC (RATIONALE 304): A Randomized Phase 3 Trial. J Thorac Oncol. 2021 Sep;16(9):1512-1522. doi: 10.1016/j.jtho.2021.05.005. Epub 2021 May 23. PMID 34033975
- [Derived] Lu S, Wang J, Yu Y, Yu X, Hu Y, Wangjun L, Li X, Liu Y, Li W, Qu X, Bao Y, Wang M. First-Line Tislelizumab Plus Chemotherapy in Advanced Non-Squamous Non-Small Cell Lung Cancer: PD-L1 >/= 50% Subgroup Analysis from the RATIONALE-304 Trial. Oncol Ther. 2025 Dec;13(4):1087-1104. doi: 10.1007/s40487-025-00378-8. Epub 2025 Sep 14. PMID 40946254
- [Derived] Lu S, Yu Y, Barnes G, Qiu X, Bao Y, Tang B. Examining the Impact of Tislelizumab Added to Chemotherapy on Health-Related Quality-of-Life Outcomes in Previously Untreated Patients With Nonsquamous Non-Small Cell Lung Cancer. Cancer J. 2022 Mar-Apr 01;28(2):96-104. doi: 10.1097/PPO.0000000000000583. PMID 35333492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 47 study centers in China.
Period: Overall Study
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Started | 223 | 111
Randomized But Not Treated | 1 | 1
Completed | 0 | 0
Not Completed | 223 | 111
Not completed — Death | 144 | 69
Not completed — Sponsor decision | 53 | 19
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Lost to Follow-up | 7 | 9
Not completed — Transferred to long term extension study | 11 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all randomized participants
Groups:
- Tislelizumab + Platinum + Pemetrexed: Tislelizumab 200 mg administered IV once every 3 weeks plus cisplatin 75 mg/m^2 or carboplatin AUC 5 once every 3 weeks for 4 to 6 cycles and pemetrexed 500 mg/m^2 once every 3 weeks until unacceptable toxicity or disease progression (each cycle is 21 days)
- Total: Total of all reporting groups
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed | Total
Number analyzed (Participants) | 223 | 111 | 334
Age, Continuous [Median (Full Range); unit: Years] | 61.0 [28 to 76] | 62.0 [25 to 75] | 61.0 [25 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 32 | 87
  Male | 168 | 79 | 247
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 223 | 111 | 334
  Not Hispanic or Latino | 223 | 111 | 334
Smoking Status [Count of Participants; unit: Participants]
  Never | 76 | 45 | 121
  Current | 32 | 13 | 45
  Former | 115 | 53 | 168
PD-L1 Expression in Tumor Cells [Count of Participants; unit: Participants] — Population: PD-L1 unevaluable refers to the participants without sample collection, not evaluable at baseline, or scored with unqualified sample.
  Participants
    <1% | 91 | 48 | 139
    1%-49% | 53 | 27 | 80
    ≥ 50% | 74 | 36 | 110
    Unevaluable | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Assessed by Independent Review Committee (IRC) Assessment
Description: PFS is defined as the time from randomization until first documentation of progression or death from any cause, whichever occurs first, as assessed by the IRC per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Time Frame: Through primary analysis data cut-off date of 23JAN2020 (up to approximately 1 year and 6 months)
Population: ITT analysis set included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 223 | 111
Months | 9.7 [7.72 to 11.53] | 7.6 [5.55 to 8.02]
Statistical Analysis 1: Comparison: Tislelizumab + Platinum + Pemetrexed vs Platinum + Pemetrexed; Test type: Superiority; p = 0.0054, One-sided, Log Rank Test; Hazard Ratio (HR) = 0.651, 95% CI 2-sided [0.465 to 0.912] — Stratified by stratification factors: disease stage (IIIB or IV) and the level of PD-L1 expression in tumor cells (>=50%, 1% to 49%, <1%)

2. Secondary Outcome: Objective Response Rate (ORR) by IRC Assessment
Description: ORR is defined as the percentage of participants with complete response (CR) or partial response (PR), as assessed by the IRC using RECIST v1.1.
Time Frame: Through study completion data cut-off date of 26APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 223 | 111
Percentage of participants | 57.8 [51.1 to 64.4] | 36.9 [28.0 to 46.6]

3. Secondary Outcome: Duration of Response (DOR) by IRC Assessment
Description: DOR is defined as the time from the first occurrence of a documented objective response to the time of documented disease progression, or death from any cause, whichever comes first, as assessed by the IRC using RECIST v1.1 in participants with documented objective responses
Time Frame: Through study completion data cut-off date of 26APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 129 | 41
Months | 10.6 [8.38 to 17.64] | 7.0 [4.99 to 10.61]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization until the date of death due to any cause
Time Frame: Through study completion data cut-off date of 26APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 223 | 111
Months | 21.4 [17.91 to 25.40] | 20.1 [14.88 to 28.12]

5. Secondary Outcome: PFS by Investigator Assessment
Description: PFS is defined as the time from randomization until first objectively documented disease progression, or death from any cause, whichever occurs first, as assessed by the investigator per RECIST v1.1
Time Frame: Through study completion data cut-off date of 26APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 223 | 111
Months | 9.7 [7.66 to 11.70] | 5.6 [4.80 to 7.66]

6. Secondary Outcome: ORR by Investigator Assessment
Description: ORR is defined as the percentage of participants with CR or PR, as assessed by the investigator using RECIST v1.1
Time Frame: Through study completion data cut-off date of 26APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 223 | 111
Percentage of participants | 57.4 [50.6 to 64.0] | 36.0 [27.1 to 45.7]

7. Secondary Outcome: DOR by Investigator Assessment
Description: DOR is defined as the time from the first occurrence of a documented objective response to the time of documented disease progression, or death from any cause, whichever comes first, as assessed by the investigator using RECIST v1.1 in participants with documented objective responses
Time Frame: Through study completion data cut-off date of 26APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 128 | 40
Months | 14.5 [9.72 to 18.66] | 8.4 [5.55 to 10.38]

8. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer (EORTC QLQ-LC13)
Description: Change from baseline in EORTC QLQ-CL13 scores for coughing, dyspnea, and chest pain . The EORTC QLQ-LC13 is a questionnaire that measures lung cancer-specific disease and treatment symptoms. It includes questions about specific symptoms in which participants respond based on a 4-point scale, where 1 is "not at all" and 4 is "very much". Raw scores are transformed into a 0 to 100 scale via linear transformation. A lower score indicates an improvement in symptoms.
Time Frame: Baseline to Cycle 5 (each cycle is 21 days)
Population: Health-related quality of life (HRQoL) analysis set included all randomized participants who received at least 1 dose of study drug and completed at least 1 HRQoL assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 222 | 110
Score on a scale
  Coughing | -13.0 [-16.6 to -9.4] | -10.8 [-15.7 to -5.9]
  Dyspnea | -1.4 [-3.5 to 0.6] | -0.3 [-3.2 to 2.6]
  Chest Pain | -7.4 [-10.4 to -4.5] | -4.2 [-8.3 to -0.2]
Statistical Analysis 1: Comparison: Tislelizumab + Platinum + Pemetrexed vs Platinum + Pemetrexed; Least squares mean difference in coughing score; Test type: Other; Least squares mean difference = -2.2, 95% CI 2-sided [-7.4 to 3.1] — Based on a constrained longitudinal data analysis model with QLQ-LC13 coughing score on the response variable and treatment by study visit interaction and randomization stratification factors as covariates
Statistical Analysis 2: Comparison: Tislelizumab + Platinum + Pemetrexed vs Platinum + Pemetrexed; Least squares mean difference in dyspnea score; Test type: Other; Least squares mean difference = -1.2, 95% CI 2-sided [-4.4 to 2.1] — Based on a constrained longitudinal data analysis model with QLQ-LC13 dyspnea score on the response variable and treatment by study visit interaction and randomization stratification factors as covariates
Statistical Analysis 3: Comparison: Tislelizumab + Platinum + Pemetrexed vs Platinum + Pemetrexed; Least squares mean difference in chest pain score; Test type: Other; Least squares mean difference = -3.2, 95% CI 2-sided [-7.6 to 1.2] — Based on a constrained longitudinal data analysis model with QLQ-LC13 chest pain score on the response variable and treatment by study visit interaction and randomization stratification factors as covariates

9. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status
Description: Change from baseline in EORTC QLQ-C30 Global Health Status/Quality of Life score. The EORTC QLQ-C30 v3.0 is a questionnaire that assesses quality of life of participants with cancer. It includes global health status and quality of life questions related to overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. A higher score indicates better health outcomes.
Time Frame: Baseline to Cycle 5 (each cycle is 21 days)
Population: HRQoL analysis set included all randomized participants who received at least 1 dose of study drug and completed at least 1 HRQoL assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 222 | 110
Score on a scale | 0.9 [-2.0 to 3.8] | -3.0 [-7.3 to 1.2]
Statistical Analysis 1: Comparison: Tislelizumab + Platinum + Pemetrexed vs Platinum + Pemetrexed; Least squares mean difference in Global Health Status/Quality of Life score; Test type: Other; Least squares mean difference = 3.9, 95% CI 2-sided [-0.9 to 8.7] — Based on a constrained longitudinal data analysis model with QLQ-LC30 Global Health Status/Quality of Life score on the response variable and treatment by study visit interaction and randomization stratification factors as covariates

10. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), which includes laboratory tests, physical exams, electrocardiogram results and vital signs, according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Time Frame: Through study completion data cut-off date of 26APR2023 (up to approximately 4 years and 9 months)
Population: Safety analysis set included all randomized participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 222 | 110
Participants
  At least one TEAE | 222 | 109
  At least one SAE | 99 | 25

11. Secondary Outcome: PFS by IRC Based on Programmed Death Ligand 1 (PD-L1) Expression
Description: PFS is defined as the time from randomization until first documentation of progression or death from any cause, whichever occurs first, as assessed by the IRC per RECIST v1.1, based on PD-L1 expression in tumor cells
Time Frame: Through study completion data cut-off date of 26APR2023 (up to approximately 4 years and 9 months)
Population: ITT analysis set included all randomized participants; participants evaluable for PD-L expression were included
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed
Number analyzed (Participants) | 218 | 111
Months
  <1% of tumor cells: number analyzed (Participants) | 91 | 48
  <1% of tumor cells | 7.6 [5.0 to 9.7] | 7.6 [4.3 to 7.9]
  1% to 49% of tumor cells: number analyzed (Participants) | 53 | 27
  1% to 49% of tumor cells | 9.7 [6.9 to 11.7] | 9.7 [5.6 to 16.8]
  ≥ 50% of tumor cells: number analyzed (Participants) | 74 | 36
  ≥ 50% of tumor cells | 17.2 [11.5 to 31.4] | 4.6 [3.5 to 9.7]

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days after the last dose of study drug; through study completion data cut-off date of 26APR2023 (up to approximately 4 years and 9 months)
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events includes all randomized participants who received ≥ 1 dose of any study treatment
Groups:
- Platinum + Pemetrexed Alone: Cisplatin 75 mg/m^2 or carboplatin AUC 5 once every 3 weeks for 4 to 6 cycles and pemetrexed 500 mg/m^2 administered IV once every 3 weeks until unacceptable toxicity or disease progression (each cycle is 21 days)
Arm/Group | Tislelizumab + Platinum + Pemetrexed | Platinum + Pemetrexed Alone
All-Cause Mortality (participants affected / at risk) | 144/223 | 69/111
Serious Adverse Events (participants affected / at risk) | 99/222 | 25/110
Other Adverse Events (participants affected / at risk) | 222/222 | 109/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Platinum + Pemetrexed (N=222) | Platinum + Pemetrexed Alone (N=110)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 2 (2) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 0 (0)
Cataract cortical (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Immune-mediated gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 3 (3)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 16 (18) | 6 (6)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 5 (5) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (3) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 2 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Platinum + Pemetrexed (N=222) | Platinum + Pemetrexed Alone (N=110)
Anaemia (Blood and lymphatic system disorders) | 185 (578) | 84 (182)
Leukopenia (Blood and lymphatic system disorders) | 65 (209) | 31 (93)
Lymphopenia (Blood and lymphatic system disorders) | 7 (9) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 84 (383) | 38 (133)
Thrombocytopenia (Blood and lymphatic system disorders) | 61 (138) | 30 (67)
Palpitations (Cardiac disorders) | 8 (8) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 11 (22) | 2 (3)
Supraventricular extrasystoles (Cardiac disorders) | 7 (15) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 12 (17) | 2 (2)
Hypothyroidism (Endocrine disorders) | 28 (45) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 8 (10) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 9 (9) | 2 (2)
Constipation (Gastrointestinal disorders) | 57 (116) | 26 (36)
Diarrhoea (Gastrointestinal disorders) | 31 (43) | 15 (20)
Mouth ulceration (Gastrointestinal disorders) | 8 (10) | 2 (2)
Nausea (Gastrointestinal disorders) | 101 (332) | 46 (86)
Toothache (Gastrointestinal disorders) | 11 (13) | 5 (6)
Vomiting (Gastrointestinal disorders) | 62 (137) | 26 (41)
Asthenia (General disorders) | 44 (68) | 17 (22)
Chest discomfort (General disorders) | 3 (3) | 6 (6)
Fatigue (General disorders) | 11 (14) | 4 (4)
Influenza like illness (General disorders) | 12 (14) | 3 (3)
Malaise (General disorders) | 42 (97) | 22 (40)
Non-cardiac chest pain (General disorders) | 14 (14) | 4 (4)
Oedema peripheral (General disorders) | 19 (21) | 6 (9)
Pyrexia (General disorders) | 40 (51) | 11 (12)
COVID-19 (Infections and infestations) | 7 (7) | 0 (0)
Pneumonia (Infections and infestations) | 19 (20) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 21 (23) | 6 (7)
Urinary tract infection (Infections and infestations) | 10 (11) | 0 (0)
Alanine aminotransferase increased (Investigations) | 116 (296) | 51 (103)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 12 (19) | 5 (8)
Aspartate aminotransferase increased (Investigations) | 104 (279) | 52 (110)
Bilirubin conjugated increased (Investigations) | 12 (18) | 1 (1)
Blood albumin decreased (Investigations) | 3 (6) | 6 (8)
Blood alkaline phosphatase increased (Investigations) | 27 (58) | 13 (17)
Blood bilirubin increased (Investigations) | 30 (57) | 10 (11)
Blood creatine phosphokinase MB increased (Investigations) | 12 (18) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 18 (29) | 5 (7)
Blood creatinine increased (Investigations) | 46 (90) | 5 (7)
Blood fibrinogen increased (Investigations) | 2 (6) | 6 (7)
Blood glucose increased (Investigations) | 15 (21) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 42 (88) | 16 (26)
Blood sodium decreased (Investigations) | 1 (1) | 4 (4)
Blood thyroid stimulating hormone increased (Investigations) | 12 (16) | 3 (7)
Blood urea increased (Investigations) | 9 (14) | 2 (2)
Blood uric acid increased (Investigations) | 5 (9) | 4 (5)
Electrocardiogram QT prolonged (Investigations) | 7 (26) | 2 (2)
Fibrin D dimer increased (Investigations) | 7 (8) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 34 (65) | 18 (25)
Haemoglobin decreased (Investigations) | 12 (30) | 8 (11)
Lymphocyte count decreased (Investigations) | 29 (88) | 6 (18)
Neutrophil count decreased (Investigations) | 149 (675) | 55 (178)
Platelet count decreased (Investigations) | 121 (381) | 46 (105)
Protein total decreased (Investigations) | 4 (6) | 4 (4)
Red blood cell count decreased (Investigations) | 7 (14) | 4 (6)
Weight decreased (Investigations) | 31 (38) | 12 (12)
Weight increased (Investigations) | 23 (29) | 4 (4)
White blood cell count decreased (Investigations) | 160 (715) | 62 (195)
Decreased appetite (Metabolism and nutrition disorders) | 81 (141) | 36 (66)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (8) | 6 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 32 (82) | 15 (20)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (10) | 6 (13)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7 (12) | 4 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 17 (36) | 10 (19)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 44 (85) | 11 (27)
Hypocalcaemia (Metabolism and nutrition disorders) | 18 (24) | 7 (7)
Hypochloraemia (Metabolism and nutrition disorders) | 16 (25) | 4 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 27 (33) | 5 (7)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (23) | 2 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 35 (59) | 14 (21)
Hypophosphataemia (Metabolism and nutrition disorders) | 8 (18) | 5 (7)
Hypoproteinaemia (Metabolism and nutrition disorders) | 19 (23) | 4 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (22) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 29 (30) | 9 (9)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 (23) | 8 (9)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 4 (4)
Dizziness (Nervous system disorders) | 31 (39) | 7 (9)
Headache (Nervous system disorders) | 13 (17) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 7 (9) | 2 (2)
Insomnia (Psychiatric disorders) | 27 (35) | 16 (17)
Proteinuria (Renal and urinary disorders) | 8 (12) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (42) | 10 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (30) | 7 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17 (23) | 9 (11)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 4 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 25 (27) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (26) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (17) | 2 (4)
Rash (Skin and subcutaneous tissue disorders) | 39 (56) | 13 (15)
Hypertension (Vascular disorders) | 7 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT03663205/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03663205/SAP_001.pdf